CLINICAL TRIAL: NCT03408730
Title: A Double-blind Randomized Controlled Trial to Assess the Lot-to-lot Consistency of Sci-B-Vac™ in Adults (CONSTANT)
Brief Title: Lot-to-lot Consistency of Sci-B-Vac™ in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VBI Vaccines Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Sci-B-Vac-002; 2017-001820-22 (EudraCT Number)
Record Dates: First submitted 2017-11-23; First posted 2018-01-24 (Actual); Results first posted 2020-10-14 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Hepatitis B Vaccines
Keywords: Hepatitis B Vaccines
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Intervention Model Description: Double-blind Randomized Controlled Trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Sci-B-Vac Lot A Hep B Vaccination (Experimental): Sci-B-Vac Lot A Hepatitis B Vaccination
  Interventions: Biological: Hepatitis B Vaccination
- Sci-B-Vac Lot B Hep B Vaccination (Experimental): Sci-B-Vac Lot B Hepatitis B Vaccination
  Interventions: Biological: Hepatitis B Vaccination
- Sci-B-Vac Lot C Hep B Vaccination (Experimental): Sci-B-Vac Lot C Hepatitis B Vaccination
  Interventions: Biological: Hepatitis B Vaccination
- Comparator: ENGERIX-B Hep B Vaccination (Active Comparator): Active Comparator: ENGERIX-B Hepatitis B Vaccination
  Interventions: Biological: Hepatitis B Vaccination

INTERVENTIONS:
Biological: Hepatitis B Vaccination — Hepatitis B Vaccination

SUMMARY:
A Controlled Trial to Assess the Lot-to-lot Consistency of Sci-B-Vac™ in Adults

DETAILED DESCRIPTION:
The primary objective of the study is to verify that the manufacturing equivalence of Sci-B-Vac™ is consistent and to compare the immunogenicity and safety of a three-dose regimen of Sci-B-Vac™ to a three-dose regimen of Engerix-B® in adults.

ELIGIBILITY:
Inclusion Criteria:

* Any gender
* Age 18-45 years
* Healthy, as determined by a physical examination and values of laboratory tests
* If female, either is not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy), is of childbearing potential and must agree to use an adequate birth control method
* Able and willing to give informed consent

Exclusion Criteria:

* Previous vaccination with any Hep B vaccine (HBV) (licensed or experimental)
* Treatment by immunosuppressant within 30 days of enrollment
* History of immunological function impairment
* Pregnancy or breastfeeding
* Immunization with attenuated vaccines (e.g. MMR) within 4 weeks prior to enrollment
* Immunization with inactivated vaccines (e.g. influenza) within 2 week prior to enrolment
* Has received blood products or immunoglobulin within 90 days of enrollment or is likely to require blood products during the study period
* Subject in another clinical trial with an investigational drug or a biologic within 30 days of enrollment
* Has received granulocyte-macrophage colony stimulating factor (G/GM-CSF) or erythropoietin (EPO) within 30 days of enrollment or likely to require GM-CSF or erythropoietin during the study period
* Any history of cancer requiring chemotherapy or radiation within 5 years of randomization or current disease.
* Any skin abnormality or tattoo that would limit post-vaccination injection site assessment
* History of allergic reactions or anaphylactic reaction to any vaccine component
* Unwilling, or unable in the opinion of the investigator, to comply with study requirements
* Immediate family members of study center staff
* Current or past hepatitis B infection or prior vaccination as evidenced by HBV markers
* Known hepatitis C infection or positive Hepatitis C serology at screening, unless treated and cured
* Known human immunodeficiency virus (HIV) infection or positive HIV serology at screening
* Renal impairment with Glomerular Filtration Rate (GFR) <90 mL/min/ 1.73 m2 at screening
* BMI ≥ 35
* Uncontrolled hypertension
* Diagnosis of Type 1 or Type 2 diabetes or HbA1C ≥ 6.5% at screening
* Any laboratory test abnormality that would be considered of Grade 1 severity or above as per FDA guidelines for grading clinical laboratory abnormalities and is considered as clinically significant by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2838 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Diaz-Mitoma, MD, PhD, Study Director — VBI Vaccines
Locations (26):
- United States (15):
  - Accel Research Sites, Birmingham, Alabama
  - Clinical Research Consortium Arizona, LLC, Tempe, Arizona
  - Anaheim Clinical Trials, Anaheim, California
  - Ruane Clinical Research Group Inc, Los Angeles, California
  - CareOne Research, North Hollywood, California
  - Avail Clinical Research, DeLand, Florida
  - Suncoast Research Group, Miami, Florida
  - Clinical Research Altanta, Atlanta, Georgia
  - Advanced Clinical Research (ACR), Boise, Idaho
  - Montana Medical Research, LLC, Missoula, Montana
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - Rapid Medical Research, Cleveland, Ohio
  - Aventiv Research Inc, Columbus, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Advanced Clinical Research (ACR), Salt Lake City, Utah
- Universitair Ziekenhuis Gent, Ghent, Oost-Vlaanderen, Belgium
- Canada (4):
  - Medicore Research Inc, Greater Sudbury, Ontario
  - Manna Toronto, Toronto, Ontario
  - Manna Montreal, Montreal, Quebec
  - Manna Research Quebec, Québec, Quebec
- University of Tampere, Tampere, Finland
- Medizinishe Hochschule Hannover, Hanover, Germany
- United Kingdom (4):
  - Oxford University, Oxford, Oxfordshire
  - Bristol Royal Hospital for Children, Bristol
  - St. George's University Hospital NHS Foundation Trust, London
  - Southampton General Hospital, Southampton

REFERENCES:
- [Derived] Vesikari T, Finn A, van Damme P, Leroux-Roels I, Leroux-Roels G, Segall N, Toma A, Vallieres G, Aronson R, Reich D, Arora S, Ruane PJ, Cone CL, Manns M, Cosgrove C, Faust SN, Ramasamy MN, Machluf N, Spaans JN, Yassin-Rajkumar B, Anderson D, Popovic V, Diaz-Mitoma F; CONSTANT Study Group. Immunogenicity and Safety of a 3-Antigen Hepatitis B Vaccine vs a Single-Antigen Hepatitis B Vaccine: A Phase 3 Randomized Clinical Trial. JAMA Netw Open. 2021 Oct 1;4(10):e2128652. doi: 10.1001/jamanetworkopen.2021.28652. PMID 34636914

RESULTS

PARTICIPANT FLOW:
Groups:
- Comparator: ENGERIX-B Hep B Vaccination: Active Comparator: ENGERIX-B Hepatitis B Vaccination
  Engerix-B® Hepatitis B Vaccination, 20ug, intramuscular (IM) injection at Days 0, 28, and 168.
- Sci-B-Vac Lot A Hep B Vaccination: Sci-B-Vac Lot A Hepatitis B Vaccination
  Sci-B-Vac® Hepatitis B Vaccination, 10ug, intramuscular (IM) injection at Days 0, 28, and 168.
- Sci-B-Vac Lot B Hep B Vaccination: Sci-B-Vac Lot B Hepatitis B Vaccination
  Sci-B-Vac® Hepatitis B Vaccination, 10ug, intramuscular (IM) injection at Days 0, 28, and 168.
- Sci-B-Vac Lot C Hep B Vaccination: Sci-B-Vac Lot C Hepatitis B Vaccination
  Sci-B-Vac® Hepatitis B Vaccination, 10ug, intramuscular (IM) injection at Days 0, 28, and 168.
Period: Overall Study
Arm/Group | Comparator: ENGERIX-B Hep B Vaccination | Sci-B-Vac Lot A Hep B Vaccination | Sci-B-Vac Lot B Hep B Vaccination | Sci-B-Vac Lot C Hep B Vaccination
Started | 712 | 711 | 709 | 706
Completed | 643 | 636 | 637 | 625
Not Completed | 69 | 75 | 72 | 81

BASELINE CHARACTERISTICS:
Population: Two subjects randomized to receive Sci-B-Vac®, one in the Lot B group and one in the Lot C group, discontinued the study before receiving any vaccinations. One of these subjects withdrew consent and the other was discontinued due to non-compliance. Data from these two subjects are not included in the Baseline Characteristics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Comparator: ENGERIX-B Hep B Vaccination | Sci-B-Vac Lot A Hep B Vaccination | Sci-B-Vac Lot B Hep B Vaccination | Sci-B-Vac Lot C Hep B Vaccination | Total
Number analyzed (Participants) | 712 | 711 | 708 | 705 | 2836
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.4 (8.10) | 33.8 (7.96) | 32.9 (8.00) | 33.9 (7.91) | 33.5 (8.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 421 | 408 | 395 | 414 | 1638
  Male | 291 | 303 | 313 | 291 | 1198
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 74 | 64 | 70 | 61 | 269
  Not Hispanic or Latino | 636 | 643 | 638 | 643 | 2560
  Unknown or Not Reported | 2 | 4 | 0 | 1 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 654 | 650 | 641 | 650 | 2595
  Race: Asian | 9 | 9 | 15 | 13 | 46
  Race: Black or African American | 38 | 46 | 43 | 34 | 161
  Race: American Indian or Alaska Native | 2 | 2 | 1 | 3 | 8
  Race: Other | 9 | 4 | 8 | 5 | 26
Region of Enrollment [Number; unit: participants]
  Canada | 31 | 31 | 29 | 30 | 121
  United States | 188 | 191 | 186 | 185 | 750
  Europe | 493 | 489 | 493 | 490 | 1965
BMI category [Count of Participants; unit: Participants]
  >30 kg/m^2 | 117 | 135 | 117 | 135 | 504
  <=30 kg/ m^2 | 595 | 576 | 591 | 570 | 2332
Smoking status [Count of Participants; unit: Participants] — Population: The smoking status of one subject in group "Sci-B-Vac Lot C Hep B Vaccination" was not documented.
  Participants
    number analyzed (Participants) | 712 | 711 | 708 | 704 | 2835
    Current smoker/ tobacco user | 136 | 139 | 142 | 125 | 542
    Former smoker/ tobacco user | 141 | 137 | 131 | 136 | 545
    Nonsmoker/ non-tobacco user | 435 | 435 | 435 | 443 | 1748

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Concentration (GMC) of Anti-HBs at Day 196 for Lot-to-Lot Consistency (Per Protocol Set 1)
Description: To demonstrate the manufacturing equivalence, in terms of immunogenicity, as measured by GMC of antibodies, of 3 independent consecutive lots of the Sci-B-Vac® 4 weeks after the third vaccination. Lot-to-lot manufacturing consistency of Sci-B-Vac® is demonstrated if the 95% CIs of the adjusted anti-HBs GMC ratios between lots are within the pre-specified range of [0.67, 1.5].
Time Frame: 4 weeks after third vaccination (Study Day 196)
Population: Per Protocol Set 1 included all subjects in the full analysis set who received all 3 vaccinations, had an evaluable serum immunogenicity samples at baseline and at the time point of interest, were seronegative at baseline, and had no major protocol violations leading to exclusion
Measure: Mean (Standard Deviation); unit: mIU/ml
Arm/Group | Sci-B-Vac Lot A Hep B Vaccination | Sci-B-Vac Lot B Hep B Vaccination | Sci-B-Vac Lot C Hep B Vaccination
Number analyzed (Participants) | 611 | 610 | 619
mIU/ml | 5883.93 (5.423) | 4824.06 (6.293) | 5505.98 (5.975)

2. Secondary Outcome: Seroprotection Rate (SPR) of Anti-HBs at Day 196 for Sci-B-Vac® Compared to Day 196 for Engerix-B® (Per Protocol Set 2)
Description: The difference in proportions [SPR(Sci-B-Vac®)-SPR(Engerix-B®)] and two-sided 95% CIs were summarized. If the lower bound of the 95% CI was > 5%, Sci-B-Vac® was to be declared non-inferior to Engerix-B®
Time Frame: 4 weeks after third vaccination (Study Day 196)
Population: Per Protocol Set 2 included all subjects in Per Protocol Set 1 excluding subjects who attended visits outside of windows including Visit 3/Day 168 (±28 days) and Visit 44/Day 196 (-7/+14 days)
Measure: Count of Participants; unit: Participants
Groups:
- Pooled Sci-B-Vac®: Pooled Sci-B-Vac Lot A, B and C Hepatitis B Vaccination
  Sci-B-Vac® Hepatitis B Vaccination, 10ug, intramuscular (IM) injection at Days 0, 28, and 168.
Arm/Group | Comparator: ENGERIX-B Hep B Vaccination | Pooled Sci-B-Vac®
Number analyzed (Participants) | 592 | 1753
Participants | 561 | 1740

3. Secondary Outcome: Percentage of Subject-reporting Solicited Local and Systemic Adverse Events (AEs)
Description: Analysis of local and systemic solicited adverse events with an interval of onset of Day 1 to Day 7 after any vaccination with either Sci-B-Vac® or Engerix-B®, in adults ≥18 years old.
Time Frame: Day of vaccine administration and six subsequent days
Population: Safety Set included all subjects in the All Enrolled Set who received at least 1 vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Comparator: ENGERIX-B Hep B Vaccination | Sci-B-Vac Lot A Hep B Vaccination | Sci-B-Vac Lot B Hep B Vaccination | Sci-B-Vac Lot C Hep B Vaccination
Number analyzed (Participants) | 712 | 711 | 708 | 705
Participants
  Pain | 384 | 527 | 536 | 542
  Tenderness | 391 | 519 | 535 | 541
  Pruritis/itching | 88 | 84 | 105 | 92
  Redness/erythema | 12 | 27 | 20 | 14
  Swelling/edema | 6 | 18 | 15 | 22
  Nausea/vomiting | 86 | 85 | 87 | 79
  Diarrhea | 105 | 94 | 87 | 96
  Headache | 268 | 255 | 275 | 281
  Fatigue | 284 | 266 | 296 | 290
  Myalgia | 231 | 289 | 316 | 337

ADVERSE EVENTS:
Time Frame: 1 year
Description: Number (%) of subject-reporting unsolicited adverse events (AEs) and serious adverse events (SAEs).
Arm/Group | Comparator: ENGERIX-B Hep B Vaccination | Sci-B-Vac Lot A Hep B Vaccination | Sci-B-Vac Lot B Hep B Vaccination | Sci-B-Vac Lot C Hep B Vaccination
All-Cause Mortality (participants affected / at risk) | 0/712 | 1/711 | 0/708 | 0/705
Serious Adverse Events (participants affected / at risk) | 3/712 | 12/711 | 18/708 | 12/705
Other Adverse Events (participants affected / at risk) | 381/712 | 376/711 | 392/708 | 399/705
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Comparator: ENGERIX-B Hep B Vaccination (N=712) | Sci-B-Vac Lot A Hep B Vaccination (N=711) | Sci-B-Vac Lot B Hep B Vaccination (N=708) | Sci-B-Vac Lot C Hep B Vaccination (N=705)
Appendicitis (Infections and infestations) | 0 | 1 | 1 | 1
Intervertebral disc protusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0 | 1
Chlamydial infection (Infections and infestations) | 0 | 0 | 0 | 1
Infectious mononucleosis (Infections and infestations) | 0 | 0 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0
Vestibular neuronitis (Infections and infestations) | 0 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Alcoholic liver disease (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Sudden cardiac death (General disorders) | 0 | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Comparator: ENGERIX-B Hep B Vaccination (N=712) | Sci-B-Vac Lot A Hep B Vaccination (N=711) | Sci-B-Vac Lot B Hep B Vaccination (N=708) | Sci-B-Vac Lot C Hep B Vaccination (N=705)
Upper respiratory tract infection (Infections and infestations) | 68 | 68 | 77 | 77
Nasopharyngitis (Infections and infestations) | 55 | 39 | 42 | 53
Influenza (Infections and infestations) | 19 | 15 | 13 | 14
Sinusitis (Infections and infestations) | 9 | 18 | 10 | 12
Urinary tract infection (Infections and infestations) | 12 | 10 | 6 | 11
Gastroenteritis (Infections and infestations) | 10 | 7 | 8 | 10
Rhinitis (Infections and infestations) | 7 | 5 | 8 | 4
Headache (Nervous system disorders) | 92 | 81 | 105 | 81
Dizziness (Nervous system disorders) | 6 | 9 | 9 | 15
Back pain (Musculoskeletal and connective tissue disorders) | 18 | 20 | 20 | 27
Myalgia (Musculoskeletal and connective tissue disorders) | 21 | 19 | 19 | 22
Neck pain (Musculoskeletal and connective tissue disorders) | 9 | 7 | 14 | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 11 | 5 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 7 | 10 | 8
Muscle tightness (Musculoskeletal and connective tissue disorders) | 10 | 7 | 4 | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9 | 5 | 3 | 5
Fatigue (General disorders) | 18 | 24 | 20 | 37
Injection site pain (General disorders) | 13 | 17 | 18 | 11
Pyrexia (General disorders) | 8 | 9 | 7 | 5
Injection site bruising (General disorders) | 7 | 7 | 8 | 6
Diarrhoea (Gastrointestinal disorders) | 8 | 14 | 11 | 10
Abdominal pain upper (Gastrointestinal disorders) | 9 | 10 | 10 | 12
Toothache (Gastrointestinal disorders) | 8 | 8 | 6 | 5
Dyspepsia (Gastrointestinal disorders) | 3 | 2 | 9 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 22 | 23 | 22 | 24
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 11 | 11 | 9
Dysmenorrhoea (Reproductive system and breast disorders) | 32 | 29 | 26 | 40
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 5 | 6 | 8
Depression (Psychiatric disorders) | 6 | 3 | 9 | 8
Anxiety (Psychiatric disorders) | 4 | 4 | 9 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-12-04): https://cdn.clinicaltrials.gov/large-docs/30/NCT03408730/SAP_000.pdf
  • Study Protocol (2018-05-09): https://cdn.clinicaltrials.gov/large-docs/30/NCT03408730/Prot_001.pdf